CLINICAL TRIAL: NCT06137196
Title: Study on Risk Identification Factors for Lung Function Impairment in AIDS Patients Recovered From Severe Pneumonia
Brief Title: Risk Identification Factors for Pulmonary Function Impairment in AIDS Patients Recovered From Severe Pneumonia
Status: Recruiting | Type: Observational
Sponsor: Guangzhou 8th People's Hospital (Other)
Responsible Party: Principal Investigator, Linghua LI, Chief physician, Guangzhou 8th People's Hospital
Other Study IDs: 202326263
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: AIDS; Pneumonia
Keywords: AIDS; Severe pneumonia; Lung function; Predictive factors
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Screening for risk factors related to lung function impairment in patients who have recovered from AIDS with severe pneumonia, to provide clinical evidence for early identification and intervention of lung function damage in this population.

DETAILED DESCRIPTION:
This is a prospective, single-center, non-randomized, clinical observational cohort study. It involves monitoring lung function at discharge (baseline, 0w), and at the 4th, 8th, 12th, 24th, and 48th weeks in patients recovering from severe pneumonia with AIDS. Basic demographic data, HIV RNA quantification, routine blood tests, blood biochemistry, arterial blood gas results, oxygenation index, immune function (CD3+, CD4+, CD8+ T cell counts), and imaging studies are also collected. Multifactorial logistic regression analysis is used to screen for clinical predictors of lung function decline in patients recovering from severe pneumonia

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed HIV infection;
2. Progression to the AIDS stage: CD4+ count <200 cells/µL and/or occurrence of opportunistic infections associated with AIDS;
3. Age between 18 to 65 years;
4. Meet the diagnostic criteria for severe pneumonia, with reference to the 2021 treatment guidelines for community-acquired pneumonia developed by the American Thoracic Society (ATS) and the Infectious Diseases Society of America (IDSA).

Exclusion Criteria:

1. Concurrent central nervous system lesions, severe liver disease, or cirrhosis;
2. Concurrent AIDS-related or non-related tumors;
3. Women who are pregnant or breastfeeding;
4. Presence of serious underlying diseases such as heart, lung, liver, kidney, etc.;
5. Alcohol abuse or drug use;
6. The researcher believes that the overall condition of the subject affects the evaluation and completion of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study participants come from the HIV/HBV co-infection cohort at the Guangzhou Eighth People's Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Obstructive Ventilatory Dysfunction | 12 weeks
  FEV1(Forced Expiratory Volume in One Second )to FVC (Forced Vital Capacity ) Ratio

SECONDARY OUTCOMES:
FEV1 | 12 weeks
  FEV1 decrease of ≥100 mL

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Eighth People's Hospital, Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No